CLINICAL TRIAL: NCT04015323
Title: The Efficacy of Interferential Current Treatment on Knee Osteoarthritis: A Randomized Double Blind Study That Compares the Effects of Different Carrier Frequencies
Brief Title: The Efficacy of Interferential Current Treatment on Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Benil Nesli Ata, MD, Principal Inversitagor, Ege University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 19-5.1/24
Record Dates: First submitted 2019-07-04; First posted 2019-07-10 (Actual); Last update posted 2020-07-22 (Actual); Status verified 2020-07

CONDITIONS: Knee Osteoarthritis
Keywords: interferential current; knee osteoarthritis; pain
MeSH Terms: conditions — Osteoarthritis, Knee; Pain | interventions — Electric Stimulation Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- IFC Therapy 2 kHz Arm (Experimental): Subjects in this group will receive interferential current to their knees with a carrier frequency of 2 kHz
  Interventions: Device: Interferential current
- IFC Therapy 4 kHz Arm (Experimental): Subjects in this group will receive interferential current to their knees with a carrier frequency of 4 kHz
  Interventions: Device: Interferential current
- IFC Therapy 8 kHz Arm (Experimental): Subjects in this group will receive interferential current to their knees with a carrier frequency of 8 kHz
  Interventions: Device: Interferential current

INTERVENTIONS:
Device: Interferential current — An electrotherapy current with different carrier frequencies

SUMMARY:
The effects of different carrier frequencies of interferential current on pain and function in patients with knee arthrosis will be compared

DETAILED DESCRIPTION:
60 patients with knee osteoarhthritis will be enrolled in the study. Subjects will be randomized to 3 groups. All patients will receive interferential currents to both their knees, with different carrier frequencies (2, 4 and 8 kilohertz (kHz) respectively). The effect of different types of carrier frequencies on pain, 10 meter walk test will be analysed.

ELIGIBILITY:
Inclusion Criteria:

* Age between 50-80 years
* Knee VAS pain scores ≥ 4
* Kellgren-Lawrence radiologic scores 2 and 3

Exclusion Criteria:

* History of knee surgery
* Inflammatory arthritis
* Paralysis of lower extremities
* Serious cardiovascular disease /presence of cardiac pacemaker
* Severe osteoarhthritis of lower extremity joints other than the knees
* History of newly diagnosed cancer (ın the last 6 months)
* Cognitive impairment

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2019-10-01 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
Change in pain scores according to visual analog scale (VAS) | At baseline, on the 3rd week visit (last day of interference therapy) and on the 7th week visit
  A visual analog scale value between 0-10. 0 meaning lack of pain and 10 meaning the worst pain the patient has experienced.

SECONDARY OUTCOMES:
Change in functional status levels according to Western Ontario and McMaster Universities Arhtiritis Incex (WOMAC) scale | At baseline, on the 3rd week visit (last day of interference therapy) and on the 7th week visit
  Womac scale is a questionnaire assessing patients' level of pain and functional status. Scores. Scores range from 0 to 96, 0 representing best and 96 representing worst scores. Pain, stiffness and functional limitation subscores are added up to obtain a total WOMAC score.
Change in pain status levels according to Western Ontario and McMaster Universities Arhtiritis Incex (WOMAC) scale | At baseline, on the 3rd week visit (last day of interference therapy) and on the 7th week visit
  Womac scale is a questionnaire assessing patients' level of pain and functional status. Scores. Scores range from 0 to 96, 0 representing best and 96 representing worst scores. Pain, stiffness and functional limitation subscores are added up to obtain a total WOMAC score.
Change in 10 meter walking test score | At baseline, on the 3rd week visit (last day of interference therapy) and on the 7th week visit
  This test is a measure that is used to assess walking speed in meters per second over 10 meters. It is used to determine functional mobility.
Change in the number of paracetamol tablets taken in a week | At baseline, on the 3rd week visit (last day of interference therapy) and on the 7th week visit
  Number of 500 mg tablets taken over one week will be written by subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Benil N Ata, M.D., Principal Investigator — Ege University
Locations (1):
- Ege University School of Medicine, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No